CLINICAL TRIAL: NCT00542841
Title: Modifier Genes in 21-Hydroxylase Deficiency
Brief Title: Examining Genetic Differences Among People With 21-Hydroxylase Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria I. New (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Maria I. New, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RDCRN 5607; U54RR019484 (NIH); RR019484
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: 21-hydroxylase Deficiency
Keywords: Adrenal Hyperplasia, Congenital; Steroid Biosynthesis Disorders
MeSH Terms: conditions — Congenital adrenal hyperplasia due to 21 hydroxylase deficiency; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Hydrocortisone withdrawal

INTERVENTIONS:
Procedure: Hydrocortisone withdrawal — This is considered a non-standard treatment. On Day 1, participants will receive one 10-mg pill of hydrocortisone. On Day 3, participants will receive intravenously a medicine called cosyntropin, a synthetic form of a hormone that the body makes. Participants will receive one last pill of hydrocortisone prior to the end of the study.

SUMMARY:
Congenital adrenal hyperplasia (CAH) is a genetic disorder that affects the amount of steroids that the body forms. The most common form of CAH is 21-hydroxylase deficiency (21OHD), which leads to cortisol deficiency. This, in turn, causes the development of mature masculine characteristics in newborn, prepubescent, and grown females and in prepubescent males. 21OHD is known to be caused by the mutation of a specific gene. However, symptom severity among people with 21OHD varies, and adults seem to be less affected than children. This study will examine participants' DNA to determine what other genes may affect the severity of 21OHD and may make the disease milder in adults than in children.

DETAILED DESCRIPTION:
CAH is a genetic steroidogenesis disorder. The most common form, 21OHD, leads to cortisol deficiency and, in turn, an excess of androgen, a hormone that promotes the development and maintenance of male sex characteristics. As a result of this androgen excess, prepubescent males and newborn, prepubescent, and grown females exhibit mature masculine characteristics. The symptoms and severity of 21OHD vary among individuals with the disease and in adults versus children. The reasons for these differences are not yet known. Current therapy for 21OHD consists of administration of glucocorticoids to replace cortisol and suppress excessive pituitary function. With more information about what genes or factors contribute to the severity of 21OHD, researchers may be able to better treat children and adults with the disease. This study will examine participants' DNA to determine what other genes may affect the severity of 21OHD and may make the disease milder in adults than in children.

People interested in participating in this 3-day inpatient study will first undergo a physical exam and provide a blood sample to determine eligibility. Eligible participants will be admitted to the study site in the morning on the first study day. A blood sample will be taken and participants will receive one 10-mg pill of hydrocortisone. Heart rates and blood pressures will be taken every 4 hours throughout the day. In the morning of Day 2, a blood sample will be taken and participants will be asked to urinate in the toilet. After this point and until the end of the study, participants will collect all urine in a jug. On the morning of Day 3, participants will complete urine collection and a blood sample will be taken. Participants will then receive intravenously a medicine called cosyntropin, a synthetic form of a hormone that the body makes. About 1 hour after this, participants will provide a final blood sample. Participants will receive one last pill of hydrocortisone prior to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 21OHD with two "severe" alleles, excluding the A/C656G mutation OR participant consents to genetic testing and a CYP21A2 mutation is identified
* Currently a patient at one of the participating centers
* Currently taking less than 15mg/m² hydrocortisone per day and has been for at least the past 3 months

Exclusion Criteria:

* History of adrenal crisis within 1 year prior to study entry
* Any coexisting condition requiring corticosteroid therapy (e.g., asthma, psoriasis)
* History of removal of both adrenal glands
* History of deficient pituitary gland function
* Current or past use of growth hormone therapy within 3 months prior to study entry
* Serum creatinine level greater than 2 mg/dL
* Systolic blood pressure less than 90 mm Hg
* History of critical illness or surgery that required general anesthesia within 1 month prior to study entry

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Serum 17-hydroxyprogesterone/cortisol ratio | After cosyntropin administration

SECONDARY OUTCOMES:
Many other serum and urine steroids, metabolites, and precursors | Before and after cosyntropin administration

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Auchus, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- University of Sao Paolo, São Paulo, São Paulo, Brazil